CLINICAL TRIAL: NCT03347565
Title: Neurocircuitry of Temperament and Motivated Behavior in Adolescent Eating Disorders
Brief Title: Brain Function in Adolescent Eating Disorders and Healthy Peers
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Christina Wierenga, Associate Professor, University of California, San Diego
Other Study IDs: 170664
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Eating Disorder
Keywords: adolescents, healthy controls
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adolescents with an Eating Disorder: Females between the ages of 14-17 currently diagnosed with an eating disorder (including ARFID, Anorexia Nervosa, Bulimia Nervosa, OSFED)
- Healthy Controls: Females between the ages of 14-17 with no psychiatric conditions

SUMMARY:
This study of adolescent eating disorders (ED) will examine the association of temperament-based classifications, brain activation during incentive processing, and ED symptoms at time of scan and 1 year later to better understand the neurobiology and symptoms of ED. We will recruit 150 females currently ill with an ED and 50 controls ages 14-17 to investigate how temperaments reflecting greater inhibition, impulsivity, or effortful control correspond to 1) clinical symptoms and 2) the brain's response to anticipation and outcome of salient stimuli, and 3) by collecting follow-up clinical data one year later, identify how temperament-based subtypes predict ED symptom change (e.g., clinical prediction). Data collection will rely on a technology called functional magnetic resonance imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Meet DSM-V criteria for an Eating Disorder or Never met criteria for an Eating disorder
* Medically stable
* Post-Pubertal (must have started menses, but subsequent loss of menses secondary to ED is fine).

Exclusion Criteria:

* Psychotic illness/other mental illness requiring hospitalization
* Current dependence on drugs or alcohol
* Physical conditions known to influence eating or weight (e.g, diabetes mellitus, pregnancy).
* On psychoactive medication
* Organic brain syndromes, delirium, psychotic disorders, or intellectual disability
* Neurological or medical disorders such as seizure disorder
* Any contraindication to undergoing an MRI
* Major depressive disorder
* Left handed

Ages: 14 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study is currently enrolling adolescent females between the ages of 14-17 who are right handed and who are either currently ill with an eating disorder or who have never had an eating disorder or any other mental illness
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Brain function | 1 year (fMRI Scan)
  Functional Magnetic Resonance imaging will be used to assess brain activation associated with inhibition, impulsivity, and control

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data including data dictionaries will be uploaded to NIMH per their data sharing requirements
Time Frame: within 1 year of data collection
Access Criteria: requests must be made to NIH